CLINICAL TRIAL: NCT05866601
Title: Effects on Anxiety in Physiotherapy Students After Simulation With Kirkpatric Evaluation as an Active Method for Learning the Clinical Enterview
Brief Title: Effects on Anxiety in Physiotherapy Students After Simulation as an Active Method for Learning the Clinical Enterview
Status: Completed | Type: Observational
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Profesor, Universidad Complutense de Madrid
Other Study IDs: 23/293.1
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Clinical Interview
Keywords: Medical education; nursing education; physiotherapy; empathy; anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Role Playing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Role-playing for learning the clinical interview — Thirty-one first-year physiotherapy students will carry out the role-playing methodology to learn how to take a clinical history in physiotherapy.
  Before and after the realization, they will be measured by means of a validated questionnaire in Spanish, the language in which they study, the variable of empathy and anxiety.
  Other Names: Role-plaiyng

SUMMARY:
The aim of the main study is to find out the effects on anxiety in physiotherapy students after role playing in the learning of the clinical history.

DETAILED DESCRIPTION:
Thirty-one first-year physiotherapy students will carry out the role-playing methodology to learn how to take a clinical history in physiotherapy.

Before and after the realization, they will be measured by means of a validated questionnaire in Spanish, the language in which they study, the variable of anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are studying the first year of Physiotherapy at the Complutense University of Madrid and wish to participate in the study.

Exclusion Criteria:

* Students who do not wish to participate in the study.

Ages: 20 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: First year physiotherapy students who carry out the role playing of the clinical history.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Anxiety Questionnaire called STAI before role playing | Through study completion, an average of 12 days
  This questionnaire allows the evaluation of trait anxiety (tendency to perceive stimuli as anxiogenic or not) and state anxiety (degree to which there are anxious elements in the person's environment at the time close to the evaluation). The response scale is Likert-type with 4 alternatives (in the Spanish adaptation from 0 to 3). Both state anxiety and trait anxiety have 20 items for assessment. Thus, the range of responses goes from 0 to 60, with a higher level of anxiety corresponding to a higher score. The Spanish adaptation has adequate psychometric properties. In addition, the scale can be applied in the adolescent population, as well as in university students, with evidence of reliability and validity.
Anxiety Questionnaire called STAI after role playing | Through study completion, an average of 12 days
  This questionnaire allows the evaluation of trait anxiety (tendency to perceive stimuli as anxiogenic or not) and state anxiety (degree to which there are anxious elements in the person's environment at the time close to the evaluation). The response scale is Likert-type with 4 alternatives (in the Spanish adaptation from 0 to 3). Both state anxiety and trait anxiety have 20 items for assessment. Thus, the range of responses goes from 0 to 60, with a higher level of anxiety corresponding to a higher score. The Spanish adaptation has adequate psychometric properties. In addition, the scale can be applied in the adolescent population, as well as in university students, with evidence of reliability and validity.
Jefferson scale before role playing | Through study completion, an average of 12 days
  To determine the empathy levels of nursing students, the validated Jefferson Empathy Scale for health professions students will be used. This scale consists of 20 items, each of which is assessed using a seven-point Likert-type response scale (from 1 = 'strongly disagree' to 7 = 'strongly agree'). These items are divided into three subscales: 'perspective taking' (11 items), which refers to the cognitive aspects of empathy; 'compassionate care' (6 items), which is characterised by a combination of cognitive and affective aspects of empathy; and 'putting oneself in the patient's shoes' (three items), considered the inverse of emotional distancing . Ten of these items are positively worded, while the other 10 are negatively worded and should be reversed. The total scores range from 20 to 140 points. Higher scores reflect higher levels of empathy.
Jefferson scale after role playing | Through study completion, an average of 12 days
  To determine the empathy levels of nursing students, the validated Jefferson Empathy Scale for health professions students will be used. This scale consists of 20 items, each of which is assessed using a seven-point Likert-type response scale (from 1 = 'strongly disagree' to 7 = 'strongly agree'). These items are divided into three subscales: 'perspective taking' (11 items), which refers to the cognitive aspects of empathy; 'compassionate care' (6 items), which is characterised by a combination of cognitive and affective aspects of empathy; and 'putting oneself in the patient's shoes' (three items), considered the inverse of emotional distancing . Ten of these items are positively worded, while the other 10 are negatively worded and should be reversed. The total scores range from 20 to 140 points. Higher scores reflect higher levels of empathy.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Eva María Martínez-Jiménez, Madrid, Madrid
  - Universidad Complutense de Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No